CLINICAL TRIAL: NCT04735653
Title: Support, Educate, Empower: The SEE Personalized Glaucoma Coaching Trial
Brief Title: The Support, Educate, Empower (SEE) Program
Acronym: SEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Paula Anne Newman-Casey, Assistant Professor of Ophthalmology and Visual Sciences, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HUM00188154; 1R01EY031337-01 (NIH)
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Glaucoma
Keywords: Ophthalmology; Glaucoma; Medication Adherence; Motivational Interviewing; Tailored Education; Self Management
MeSH Terms: conditions — Glaucoma; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Glaucoma Coaching (Experimental): This is a six-month personalized glaucoma coaching program where a coach trained in motivational interviewing (MI)-based counseling uses a web-based tool that generates tailored education to help glaucoma patients identify their barriers to optimal medication adherence and explore potential solutions during three in-person coaching sessions. The coach provides between-session support through four phone calls, with two phone calls between the first and second sessions and one call after each subsequent session. Participants can elect to receive any of the following types of alarm when a dose of medication is due: visual or audible alert or automated text or phone call reminder. Glaucoma medication adherence will be monitored electronically for all participants between the baseline visit and the exit visit six months later.
  Interventions: Behavioral: Personalized Glaucoma Coaching
- Enhanced standard care (Active Comparator): Participants will receive non-tailored educational materials about glaucoma from leading sources by mail every 2 months for a total of 3 mailings during the 6-month study period. Glaucoma medication adherence will be monitored electronically for all participants between the baseline visit and the exit visit six months later.
  Interventions: Behavioral: Enhanced Standard care

INTERVENTIONS:
Behavioral: Personalized Glaucoma Coaching — This is a six-month personalized glaucoma coaching program where a coach trained in motivational interviewing (MI)-based counseling uses a web based tool that generates tailored education to help glaucoma patients identify their barriers to optimal medication adherence and explore potential solutions during three in-person coaching sessions. The coach provides between-session support through four phone calls, with two phone calls between the first and second session and one phone call after each subsequent session. Participants can elect to receive any of the following type of alarm when a dose of medication is due: visual or audible alert or automated text or phone call reminder. Glaucoma medication adherence will be monitored electronically for all participants between the baseline visit and the exit visit six months later.
  Arms: Personalized Glaucoma Coaching
Behavioral: Enhanced Standard care — Participants will receive non-tailored educational materials about glaucoma from leading sources by mail every 2 months for a total of 3 mailings during the 6-month study period. Glaucoma medication adherence will be monitored electronically for all participants between the baseline visit and the exit visit six months later.
  Arms: Enhanced standard care

SUMMARY:
This study will test whether the Support, Educate, Empower (SEE) personalized Glaucoma Coaching Program improves eye drop medication adherence among glaucoma patients compared to enhanced standard care in a randomized controlled clinical trial. As a secondary outcome, the study will test whether glaucoma related distress decreases among SEE program participants compared to the control group.

The study hypothesis is that glaucoma patients with poor adherence who receive motivational-interviewing based counseling and personalized education from a trained non-physician glaucoma coach through the SEE Program will improve their medication adherence compared to glaucoma patients standard care enhanced by additional educational handouts.

ELIGIBILITY:
Inclusion Criteria:

* Taking greater or equal to 1 ocular hypotensive medication with a diagnosis of any kind of glaucoma, suspected glaucoma or ocular hypertension
* Did not opt-out from recruitment letter

Exclusion Criteria:

* Do not speak English
* Have a diagnosed serious mental illness (for example, Schizophrenia)
* Diagnosed cognitive impairment
* Do not instill their own eye drops
* Had laser or incisional glaucoma surgery within three months of enrollment or scheduled during the six-month study period
* Unable to attend all study visits
* Active ocular infection or uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Newman-Casey, MD MS, Principal Investigator — University of Michigan; Suzanne Winter, MS, Study Director — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 236 participants were consented. 235 were randomized. The unrandomized individual was determined to be ineligible post-consenting.
Groups:
- SEE Intervention - Personalized Glaucoma Coaching: SEE Intervention - Personalized Glaucoma Coaching: This is a six-month personalized glaucoma coaching program where a coach trained in motivational interviewing (MI)-based counseling uses a web based tool that generates tailored education to help glaucoma patients identify their barriers to optimal medication adherence and explore potential solutions during three in-person coaching sessions. The coach provides between-session support through four phone calls, with two phone calls between the first and second session and one phone call after each subsequent session. Participants can elect to receive any of the following type of alarm when a dose of medication is due: visual or audible alert or automated text or phone call reminder.
- Enhanced Care Control: Enhanced Care Control: Participants will receive non-tailored educational materials about glaucoma from leading sources by mail every 2 months for a total of 3 mailings during the 6-month study period.
Period: Overall Study
Arm/Group | SEE Intervention - Personalized Glaucoma Coaching | Enhanced Care Control
Started | 117 | 118
Completed (Participants who "completed" the study attended the exit visit at the end of the six month study.) | 90 | 107
Not Completed | 27 | 11
Not completed — Lost to Follow-up | 17 | 7
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Death | 0 | 2
Not completed — Removed due to determination of participant noncompliance | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SEE Intervention - Personalized Glaucoma Coaching | Enhanced Care Control | Total
Number analyzed (Participants) | 117 | 118 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (11.5) | 68.2 (10.4) | 67.3 (10.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 64 | 60 | 124
  Male | 53 | 57 | 110
  Not Reported | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 101 | 101 | 202
  Unknown or Not Reported | 14 | 13 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 68 | 71 | 139
  White | 32 | 36 | 68
  Asian | 6 | 4 | 10
  Other | 5 | 5 | 10
  Not Reported | 6 | 2 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 117 | 118 | 235

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Electronically Monitored Medication Adherence Over Six Months
Description: Medication adherence will be measured objectively using electronic monitors with a bottle-in-bottle technique where all glaucoma medications are placed inside electronic pill bottles. An adherent event is defined as using an eye drop medication within a specified time window of a dose on the previous day.
  Adherence will be calculated as the percentage of doses taken on time divided by total doses prescribed over the six-month study period. The calculation censored participants at the time of withdrawal, loss to follow-up, or disengagement (attended the exit visit but may have gone some time before this visit without adherence monitor activity) and their adherence was calculated only during the reduced time on study. Additionally, times noted where monitors malfunctioned or went unused due to vacation or hospitalization were excluded.
Time Frame: Up to 6 months
Population: Data is shown for participants who provided data for this outcome.
Measure: Mean (Standard Deviation); unit: percent adherence
Arm/Group | SEE Intervention - Personalized Glaucoma Coaching | Enhanced Care Control
Number analyzed (Participants) | 113 | 114
percent adherence | 77.6 (19.7) | 58.0 (25.2)
Statistical Analysis 1: Comparison: SEE Intervention - Personalized Glaucoma Coaching vs Enhanced Care Control; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — A Wilcoxon rank-sum test was used instead of ANOVA due to the non-normality of the adherence outcomes. We did not block on clinic due to differences in sample characteristics by site; Medication adherence was compared between groups with a Wilcoxon rank-sum test

2. Primary Outcome: Percentage of Participants Who Achieved >= 80% Medication Adherence Over the 6 Month Study Period
Description: Medication adherence will be measured objectively using electronic monitors with a bottle-in-bottle technique where all glaucoma medications are placed inside electronic pill bottles. An adherent event is defined as using an eye drop medication within a specified time window of a dose on the previous day.
  Adherence will be calculated as the percentage of doses taken on time divided by total doses prescribed over the six-month study period. The calculation censored participants at the time of withdrawal, loss to follow-up, or disengagement (attended the exit visit but may have gone some time before this visit without adherence monitor activity) and their adherence was calculated only during the reduced time on study. Additionally, times noted where monitors malfunctioned or went unused due to vacation or hospitalization were excluded.
  Continuous percentage adherence was dichotomized to a binary outcome as >= 80% vs < 80% medication adherence.
Time Frame: Up to 6 months
Population: Data is shown for participants who provided data for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | SEE Intervention - Personalized Glaucoma Coaching | Enhanced Care Control
Number analyzed (Participants) | 113 | 114
Participants
  Adherence >= 80% | 62 | 27
  Adherence < 80% | 51 | 87
Statistical Analysis 1: Comparison: SEE Intervention - Personalized Glaucoma Coaching vs Enhanced Care Control; Test type: Superiority; p < 0.001, Chi-squared — A chi-squared test was used instead of Cochran-Mantel-Haenszel test due to site differences. Site differences will be incorporated into multivariable models to investigate moderating effects with treatment on the outcome in future analyses

3. Secondary Outcome: Change in Glaucoma-related Distress
Description: Glaucoma-related Distress will be measured by the Diabetes Distress Scale adapted for glaucoma, a 17-item scale where each item is assessed on a 6-point Likert scale. A composite score is calculated as a mean of the 17 items, ranging from 1 to 6, where a higher score indicates a higher distress level. Mean change in Glaucoma-related Distress will be compared between the intervention and control groups.
  Six-month change from baseline is calculated by subtracting the baseline value from the six-month score. Negative number for change indicates that participant distress decreased over time and a positive number for change would indicate that distress increased.
Time Frame: 6 months
Population: Data is reported for people who came to the exit visit and provided both baseline and 6-month data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SEE Intervention - Personalized Glaucoma Coaching | Enhanced Care Control
Number analyzed (Participants) | 90 | 107
score on a scale
  Baseline | 2.5 (0.9) | 2.4 (0.8)
  6 months | 1.9 (0.8) | 2.2 (0.9)
  6 month change from Baseline | -0.6 (0.9) | -0.2 (0.7)
Statistical Analysis 1: Comparison: SEE Intervention - Personalized Glaucoma Coaching vs Enhanced Care Control; Test type: Superiority; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to -0.1] — Adjustment for site was not performed. Site differences will be incorporated into multivariable models to investigate moderating effects with treatment on the outcome in future analyses

ADVERSE EVENTS:
Time Frame: 6 months
Description: IOP was checked five times in the intervention group and twice in the control group.
Arm/Group | SEE Intervention - Personalized Glaucoma Coaching | Enhanced Care Control
All-Cause Mortality (participants affected / at risk) | 0/117 | 2/118
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/118
Other Adverse Events (participants affected / at risk) | 18/117 | 7/118
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEE Intervention - Personalized Glaucoma Coaching (N=117) | Enhanced Care Control (N=118)
High Intraocular Pressure (IOP) (Eye disorders) | 18 (117) | 7 (118)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT04735653/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT04735653/ICF_001.pdf